CLINICAL TRIAL: NCT05818670
Title: Comparison Between Tamsulosin and Tadalafil in Management of Benign Prostatic Hyperplasia A Randomised Trial
Brief Title: Comparison Between Tamsulosin and Tadalafil in Management of Benign Prostatic Hyperplasia Long Term Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tadalafil vs tamsulosin in bph
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: BPH
Keywords: tamsulosin; tadalafil; BPH; Randomised trial; longterm; discontinuation rate
MeSH Terms: interventions — Tamsulosin; Tadalafil

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tamsulosin (Active Comparator): patients with benign prostatic hyperplasia (BPH) and erectile dysfunction (ED) treated by tamsulosin with 12 months follow up
  Interventions: Drug: Tamsulosin
- tadalafil (Active Comparator): patients with benign prostatic hyperplasia (BPH) and erectile dysfunction (ED) treated by tadalafil 5 mg with 12 months follow up
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tamsulosin — long term follow up
  Arms: tamsulosin
Drug: Tadalafil — long term follow up
  Arms: tadalafil

SUMMARY:
Comparison between tamsulosin and Tadalafil in management of benign prostatic hyperplasia A Randomised Trial

DETAILED DESCRIPTION:
Assessment of the discontinuation rate of tamsulosin and tadalafil after 12 months follow up either and evaluate the changes in urinary parameters and sexual parameters in patients with lower urinary tract symptoms due to BPH concomitant with erectile dysfunction. We tried to overcome the limitations of the previous studies by designing a prospective randomized controlled trial as the present study is the first randomized controlled trial that evaluate the safety, discontinuation rate and efficacy of tadalafil compared with tamsulosin for long term follow up (12 months).

ELIGIBILITY:
Inclusion Criteria:

* patients with Lower Urinary Tract Symptoms
* married and sexually active
* age more than 50 years
* IPSS more than 12
* Q max less than 15 ml/s
* Post voiding residual less than 150 ml

Exclusion Criteria:

* prostatic adenocarcinoma
* cardiac patients on nitrates, patient with unstable angina or recent history of myocardial infarction
* vesical stones
* active Urinary Tract Infection
* patient refused participation in the study

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
drug discontinuation rate | 12 months
  drug discontinuation rate either : lack of response, adverse events or poor compliance

SECONDARY OUTCOMES:
changes in urinary parameters | 12 months
  detect the improvement in International Prostate Symptom Score (IPSS) . The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms
changes in uroflowmetry | 12 months
  detect the changes in maximum flow rate (Q max) as Qmax below 10 ml /sec is obstructed flow curve , between 10 to 15 ml / sec is equivocal and above 15 ml/ sec is normal
changes in post voiding residual urine | 12 months
  measured by pelvic ultrasound after micturation to detect the amount of residual urine in milliliter.
changes in sexual parameters | 12 months
  changes in International Index of Erectile Function(IIEF) . IIEF questionnaire is classified as : No erectile dysfunction (26-30points), Mild ED (score 22-25), Mild to moderate (17-21), Moderate ED (score 11-16), Severe ED (score ≤ 10)

CONTACTS AND LOCATIONS:
Overall Officials: ahmed A elqaffas, master, Principal Investigator — Mansoura urology and nephrology center (UNC)
Locations (2):
- Egypt (2):
  - Ahmed Atta Elqaffas, Al Mansurah, Dakahlia Governorate
  - Urology and Nephrology Center at Mansoura University, Al Mansurah, Dakahlia Governorate